CLINICAL TRIAL: NCT00127673
Title: Effectiveness of PTSD Treatment: CBT Versus Sertraline
Brief Title: Comparison of Two Treatments for Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Norah Feeny, Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH066347 (NIH); R01MH066348 (NIH)
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Antidepressants; Cognitive behavior therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CBT no choice (Active Comparator): Participants will receive no choice cognitive behavioral therapy (CBT no choice)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- CBT choice (Active Comparator): Participants will receive choice cognitive behavioral therapy (CBT choice)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- sertraline no choice (Active Comparator): Participants will receive no choice sertraline (sertraline no choice)
  Interventions: Drug: Sertraline
- sertraline choice (Active Comparator): Participants will receive choice sertraline (sertraline choice)
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — The dose of sertraline will be up to 200 mg daily for 10 weeks. There will also be weekly meetings with study psychiatrist.
  Other Names: Zoloft
  Arms: sertraline choice; sertraline no choice
Behavioral: Cognitive behavioral therapy (CBT) — CBT will include 10 weekly sessions of individual cognitive behavioral therapy.
  Other Names: Prolonged exposure (PE)
  Arms: CBT choice; CBT no choice

SUMMARY:
This study will compare the short- and long-term effectiveness of two different treatments for people with post-traumatic stress disorder.

DETAILED DESCRIPTION:
Exposure to traumatic events, such as automobile accidents and assault, can cause individuals to develop persistent psychological difficulties such as post-traumatic stress disorder (PTSD). PTSD is an anxiety disorder characterized by avoidance, hyperarousal symptoms, and mental re-experiencing of the traumatic event. PTSD is a serious condition that may cause social and psychological impairment; therefore, safe and effective treatments are needed. Both CBT and antidepressant therapy have been shown to effectively treat PTSD symptoms; however, comparisons of the treatments are limited. This study will compare the short- and long-term effectiveness of CBT and the antidepressant sertraline.

Participants will either be randomly assigned to CBT or sertraline, or they will be able to choose one of the two treatments, which will be given for 10 weeks, followed by 24 months of follow-up assessments. Participants in the CBT group will have 10 weekly sessions of therapy. During the therapy sessions, participants will be encouraged to confront their general fears and the memory of their trauma through repeated storytelling. Participants will also be encouraged to practice the techniques learned in therapy in everyday life. Participants in the antidepressant group will take sertraline daily for 10 weeks. These participants will be seen weekly by a psychiatrist who will offer general encouragement and support, monitor response to medication, and record any side effects participants may be experiencing. The medication may be adjusted according to a dosing schedule and based on the study doctor's judgment. At the end of 10 weeks, participants in the antidepressant group will have the choice of either tapering the medication gradually to minimize the chance of withdrawal symptoms or staying on the medication for up to 24 months. Participants who do not respond to their assigned or chosen treatment will be offered the other treatment for 10 weeks. Self-report scales and questionnaires will be used to assess participants' PTSD symptoms, depression, anxiety, and social functioning. These assessments will occur at 3, 6, 12, and 24 months after the study treatment period.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of PTSD
* Experienced traumatic event at least 12 weeks prior to study entry
* Willingness to discontinue current CBT or antidepressant treatment

Exclusion Criteria:

* Current diagnosis of schizophrenia or delusional disorder
* Medically unstable bipolar disorder, depression with psychotic features, or depression requiring psychiatric treatment
* Current diagnosis of alcohol or substance dependence within 3 months prior to study entry
* Ongoing intimate relationship with the perpetrator of the traumatic event
* History of nonresponse to either CBT or sertraline
* Medical contraindication for sertraline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah C. Feeny, PhD, Principal Investigator — Department of Psychology, Case Western Reserve University; Lori A. Zoellner, PhD, Principal Investigator — Department of Psychology, University of Washington
Locations (1):
- Department of Psychology, University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Gauthier GM, PeConga EK, Mohr JL, Feeny NC, Zoellner LA. Prospective stability of memory for peritraumatic dissociation and anxiety: Replication and extension examining PTSD treatment modality and response. Psychol Trauma. 2025 Feb;17(2):429-437. doi: 10.1037/tra0001790. Epub 2024 Nov 7. PMID 39509231
- [Derived] Rosencrans PL, Zoellner LA, Feeny NC. A network approach to posttraumatic stress disorder: Comparing interview and self-report networks. Psychol Trauma. 2024 Feb;16(2):340-346. doi: 10.1037/tra0001151. Epub 2021 Oct 21. PMID 34672659
- [Derived] Graham B, Garcia NM, Bergman HE, Feeny NC, Zoellner LA. Prolonged Exposure and Sertraline Treatments for Posttraumatic Stress Disorder Also Improve Multiple Indicators of Social Functioning. J Trauma Stress. 2020 Aug;33(4):488-499. doi: 10.1002/jts.22570. Epub 2020 Jul 13. PMID 32662191
- [Derived] Zoellner LA, Roy-Byrne PP, Mavissakalian M, Feeny NC. Doubly Randomized Preference Trial of Prolonged Exposure Versus Sertraline for Treatment of PTSD. Am J Psychiatry. 2019 Apr 1;176(4):287-296. doi: 10.1176/appi.ajp.2018.17090995. Epub 2018 Oct 19. PMID 30336702
- [Derived] Le QA, Doctor JN, Zoellner LA, Feeny NC. Effects of treatment, choice, and preference on health-related quality-of-life outcomes in patients with posttraumatic stress disorder (PTSD). Qual Life Res. 2018 Jun;27(6):1555-1562. doi: 10.1007/s11136-018-1833-4. Epub 2018 Mar 14. PMID 29541927
- [Derived] Le QA, Doctor JN, Zoellner LA, Feeny NC. Cost-effectiveness of prolonged exposure therapy versus pharmacotherapy and treatment choice in posttraumatic stress disorder (the Optimizing PTSD Treatment Trial): a doubly randomized preference trial. J Clin Psychiatry. 2014 Mar;75(3):222-30. doi: 10.4088/JCP.13m08719. PMID 24717377
- [Derived] Le QA, Doctor JN, Zoellner LA, Feeny NC. Minimal clinically important differences for the EQ-5D and QWB-SA in Post-traumatic Stress Disorder (PTSD): results from a Doubly Randomized Preference Trial (DRPT). Health Qual Life Outcomes. 2013 Apr 12;11:59. doi: 10.1186/1477-7525-11-59. PMID 23587015
- See also: Click here for more information about the effectiveness of CBT and sertraline for PTSD — http://faculty.washington.edu/zoellner/PTSDTx.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- NoChoice_CBT: Participants will receive no choice cognitive behavioral therapy
  Cognitive behavioral therapy (CBT): CBT will include 10 weekly sessions of individual cognitive behavioral therapy.
- Choice_CBT: Participants will receive choice cognitive behavioral therapy
  Cognitive behavioral therapy (CBT): CBT will include 10 weekly sessions of individual cognitive behavioral therapy.
- NoChoice_SER: Participants will receive no choice sertraline
  Sertraline: The dose of sertraline will be up to 200 mg daily for 10 weeks. There will also be weekly meetings with study psychiatrist.
- Choice_SER: Participants will receive choice sertraline
  Sertraline: The dose of sertraline will be up to 200 mg daily for 10 weeks. There will also be weekly meetings with study psychiatrist.
Period: Overall Study
Arm/Group | NoChoice_CBT | Choice_CBT | NoChoice_SER | Choice_SER
Started | 48 | 61 | 55 | 36
Completed | 23 | 44 | 35 | 25
Not Completed | 25 | 17 | 20 | 11

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | NoChoice_CBT | Choice_CBT | NoChoice_SER | Choice_SER | Total
Number analyzed (Participants) | 48 | 61 | 55 | 36 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (11.4) | 37.1 (11.3) | 38.9 (11.3) | 38.3 (11.4) | 36.60 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 46 | 43 | 25 | 152
  Male | 10 | 15 | 12 | 11 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 3 | 10
  Not Hispanic or Latino | 47 | 58 | 52 | 33 | 190
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 1 | 5
  Asian | 2 | 6 | 2 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 10 | 12 | 12 | 9 | 43
  White | 30 | 38 | 38 | 24 | 130
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 3 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms
Description: total score, range from 0-80, higher scores are more severe
Time Frame: Post-treatment, ten weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT no Choice | CBT Choice | Sertraline no Choice | Sertraline Choice
Number analyzed (Participants) | 42 | 53 | 33 | 27
units on a scale | 10.02 (10.27) | 10.87 (8.75) | 15.12 (14.03) | 10.78 (7.59)

2. Primary Outcome: Depression Symptoms
Description: Hamilton Depression Rating Scale (HAMD), total score, scoring range 0-50, with higher scores more severe depression
Time Frame: Measured at Post-Treatment, at 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT no Choice | CBT Choice | Sertraline no Choice | Sertraline Choice
Number analyzed (Participants) | 42 | 53 | 33 | 27
units on a scale | 10.33 (10.33) | 12.13 (8.67) | 15.24 (13.90) | 12.11 (10.12)

3. Primary Outcome: State Anxiety
Description: State-Trait Anxiety Inventory - State version, total score, scoring range, 0-63, with higher scores more severe
Time Frame: Measured at Post-Treatment, at 10 weeks
Population: Completer analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NoChoice_CBT | Choice_CBT | NoChoice_SER | Choice_SER
Number analyzed (Participants) | 42 | 53 | 33 | 27
units on a scale | 39.16 (13.83) | 38.79 (13.13) | 46.89 (18.91) | 38.72 (12.48)

4. Secondary Outcome: Quality of Life Functioning
Description: Sheehan Disability Scale (SDS), total score, scoring range 0-30 , higher scores indicative of worse functional impairment
Time Frame: Measured at Post-Treatment, at 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT no Choice | CBT Choice | Sertraline no Choice | Sertraline Choice
Number analyzed (Participants) | 42 | 53 | 33 | 27
units on a scale | 8.82 (6.24) | 11.68 (8.23) | 14.06 (10.38) | 10.78 (9.40)

ADVERSE EVENTS:
Time Frame: Approximately 4 months
Description: After randomization through acute treatment until post-treatment assessment
Arm/Group | NoChoice_CBT | Choice_CBT | NoChoice_SER | Choice_SER
Serious Adverse Events (participants affected / at risk) | 1/48 | 2/61 | 0/55 | 0/36
Other Adverse Events (participants affected / at risk) | 2/48 | 3/61 | 4/55 | 5/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NoChoice_CBT (N=48) | Choice_CBT (N=61) | NoChoice_SER (N=55) | Choice_SER (N=36)
Chest pain/shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney Stones (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NoChoice_CBT (N=48) | Choice_CBT (N=61) | NoChoice_SER (N=55) | Choice_SER (N=36)
Headache/dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (6)
Gastrointestinal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Delayed ejaculation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitancy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospital admission after accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral tonsilitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient increased in agitation/anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No